CLINICAL TRIAL: NCT04333576
Title: A Phase 3b Study to Evaluate the Safety and Efficacy of Elagolix in Combination With Combined Oral Contraceptives in Premenopausal Women With Documented Endometriosis and Associated Moderate to Severe Pain
Brief Title: Study Of Oral Elagolix Tablets In Combination With Combined Oral Contraceptive Capsules/Tablets To Assess Dysmenorrhea Response In Adult Female Participants With Endometriosis And Associated Moderate To Severe Pain
Acronym: ELARIS EM-COC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M18-969
Record Dates: First submitted 2020-04-02; First posted 2020-04-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Endometriosis
Keywords: Endometriosis; Elagolix; Combined oral contraceptives (COC); Orilissa; Dysmenorrhea
MeSH Terms: conditions — Endometriosis; Dysmenorrhea | interventions — elagolix; Contraceptives, Oral, Combined

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Double-Blind: Placebo (Placebo Comparator): Participants will receive double-blind placebo on Day 1 for 3 months. At month 4, participants will receive open-label elagolix in combination with COC (combined oral contraceptive) for 15 months. Participants will be followed-up for up to 12 months.
  Interventions: Drug: Elagolix; Drug: Placebo; Drug: Combined Oral Contraceptive
- Double-Blind: Elagolix (Experimental): Participants will receive double-blind Elagolix on Day 1 for 3 months. At month 4, participants will receive open-label elagolix in combination with COC (combined oral contraceptive) for 15 months. Participants will be followed-up for up to 12 months.
  Interventions: Drug: Elagolix; Drug: Combined Oral Contraceptive
- Double-Blind: Elagolix + COC (Experimental): Participants will receive double-blind elagolix in combination with COC (combined oral contraceptive) on Day 1 for 3 months. At month 4, participants will receive open-label elagolix in combination with COC for 15 months. Participants will be followed-up for up to 12 months.
  Interventions: Drug: Elagolix; Drug: Combined Oral Contraceptive

INTERVENTIONS:
Drug: Elagolix — Tablet:Oral
  Other Names: ABT-620; Orilissa
Drug: Placebo — Tablet:Oral
  Arms: Double-Blind: Placebo
Drug: Combined Oral Contraceptive — Tablet:Oral

SUMMARY:
Endometriosis is a painful disorder of the uterus affecting 6-10% of women of childbearing age. Endometriosis affects daily activities, social relationships, sexuality and sexual activity, and mental health. This study will evaluate how well elagolix in combination with combined oral contraceptives (COC) works within the body and/or how safe it is compared to placebo (does not contain treatment drug). This study will assess the dysmenorrhea (painful periods) response in participants with endometriosis and associated pain.

Elagolix is an approved drug for the management of moderate to severe pain associated with endometriosis. Participants are randomly put in 1 of 3 groups, called treatment arms. Each group receives a different treatment. There is a 1 in 3 chance that participants will be assigned to placebo. Adult female participants who still have periods with a diagnosis of endometriosis will be enrolled. Around 800 participants will be enrolled in the study at multiple sites in the United States, including Puerto Rico.

Participants will receive oral elagolix or placebo tablets in combination with combined oral contraceptive (COC) or placebo capsules for 3 months. All the participants will receive elagolix tablets in combination with COC tablets from Month 4 through Month 18.

There will be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the course of the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Documented surgical confirmation of endometriosis and associated moderate to severe pain.
* Participants must agree to use dual non-hormonal methods of contraception consistently during washout (if applicable), screening, and 3-month double-blind placebo-controlled treatment periods of the study.
* Participant, in the investigator's opinion must be an appropriate candidate to receive combined oral contraceptives (COCs).

Exclusion Criteria:

* Pregnant or breastfeeding or planning a pregnancy until completion of the study.
* Surgical history of hysterectomy or bilateral oophorectomy.
* Participant has osteoporosis or other metabolic bone disease or clinically significant gynecological findings from Screening.
* Participant has any other active chronic pain condition that would interfere with their assessment of endometriosis-related pain.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 800 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Responders Based on Dysmenorrhea (DYS) Pain Scale | Month 3
  DYS response is measured by the 4-point Endometriosis Daily Pain Impact Scale (none, mild, moderate, severe) and with stable or decreased analgesic use.

SECONDARY OUTCOMES:
Percentage of Responders Based on Non-Menstrual Pelvic Pain (NMPP) Pain Scale | Month 3
  NMPP response is measured by the 4-point Endometriosis Daily Pain Impact Scale (none, mild, moderate, severe) and with stable or decreased analgesic use.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (179):
- United States (176):
  - Pinnacle Research Group /ID# 217062, Anniston, Alabama
  - ACCEL Research Sites /ID# 218044, Birmingham, Alabama
  - Alabama Clinical Therapeutics /ID# 217166, Birmingham, Alabama
  - Alabama Clinical Therapeutics /ID# 222301, Birmingham, Alabama
  - University of Alabama at Birmingham - Women's and Infant's Center /ID# 224503, Birmingham, Alabama
  - Trinity Research Group /ID# 246932, Dothan, Alabama
  - Southern Women's Specialists PC /ID# 217143, Fairhope, Alabama
  - Women's Health Alliance of Mobile /ID# 222591, Mobile, Alabama
  - Mobile, OBGYN P.C. /ID# 217135, Mobile, Alabama
  - North Valley Women's Care /ID# 217092, Glendale, Arizona
  - MomDoc Womens Health Research /ID# 221661, Phoenix, Arizona
  - Applied Research Center of Arkansas /ID# 248494, Little Rock, Arkansas
  - Unity Health- Searcy Medical Center /ID# 217050, Searcy, Arkansas
  - Diagnamics Inc. /ID# 225385, Encinitas, California
  - Atella Clinical Research /ID# 224024, La Palma, California
  - Valley Renal Medical Group Research /ID# 228614, Northridge, California
  - Futura Research, Org /ID# 217361, Norwalk, California
  - Northern California Research /ID# 217301, Sacramento, California
  - A & B Clinical Research /ID# 224471, San Diego, California
  - Advanced Clinical Research Center, LLC /ID# 248398, San Diego, California
  - Rocky Mountain Internal Medicine - Aurora /ID# 245161, Aurora, Colorado
  - Velocity Clinical Research - Denver /ID# 217297, Denver, Colorado
  - Boeson Research - Grand Junction /ID# 248580, Grand Junction, Colorado
  - Advanced Women's Health Institute /ID# 217150, Greenwood Village, Colorado
  - Red Rocks OB/GYN /ID# 217103, Lakewood, Colorado
  - Reproductive Assoc of Delaware /ID# 227764, Newark, Delaware
  - Medstar Health Research Institute /ID# 244937, Washington D.C., District of Columbia
  - James A. Simon, MD, PC /ID# 218116, Washington D.C., District of Columbia
  - Topaz Clinical Research /ID# 218615, Apopka, Florida
  - Ideal Clinical Research Inc. /ID# 218832, Aventura, Florida
  - Helix Biomedics, LLC /ID# 218649, Boynton Beach, Florida
  - Olympian Clinical Research /ID# 244426, Clearwater, Florida
  - Women's Medical Research Group /ID# 218524, Clearwater, Florida
  - Doral Medical Research, LLC /ID# 225146, Doral, Florida
  - Universal Axon Clinical Research /ID# 248553, Doral, Florida
  - KO Clinical Research, LLC /ID# 217173, Fort Lauderdale, Florida
  - Alliance for Multispecialty Research (AMR) - Fort Myers /ID# 217061, Fort Myers, Florida
  - Solutions Through Adv Rch /ID# 220973, Jacksonville, Florida
  - Care Partners Clinical Research /ID# 217042, Jacksonville, Florida
  - Vida Clinical Research /ID# 245325, Kissimmee, Florida
  - Kissimmee Clinical Research /ID# 224749, Kissimmee, Florida
  - South Florida Wellness & Clinic /ID# 222897, Margate, Florida
  - GRE Clinical Research, LLC /ID# 246579, Miami, Florida
  - Gold Coast Health Research, LLC /ID# 248624, Miami, Florida
  - Admed Research LLC /ID# 227679, Miami, Florida
  - The Miami Research Group Inc /ID# 246578, Miami, Florida
  - Innova Pharma Research /ID# 245354, Miami, Florida
  - Ocean Blue Medical Research Center, Inc /ID# 217286, Miami Springs, Florida
  - Salom Tangir, LLC /ID# 217273, Miramar, Florida
  - Suncoast Clinical Research Pasco County /ID# 217249, New Port Richey, Florida
  - Advanced Research Institute, Inc /ID# 217206, New Port Richey, Florida
  - Segal Institute for Clinical Research /ID# 221518, North Miami, Florida
  - A Premier Medical Research of FL /ID# 216908, Orange City, Florida
  - Osceola Gynecology, LLC - Orlando /ID# 227194, Orlando, Florida
  - Omega Research Group /ID# 216907, Orlando, Florida
  - Clinical Associates of Orlando /ID# 218114, Orlando, Florida
  - Duplicate_Suncoast Clinical Research - Palm Harbor /ID# 219133, Palm Harbor, Florida
  - Royal Research,Corp /ID# 221356, Pembroke Pines, Florida
  - Physician Care Clin. Res., LLC /ID# 217264, Sarasota, Florida
  - Tampa General Hospital - Tampa - General Circle /ID# 217146, Tampa, Florida
  - GCP Clinical Research, LLC /ID# 217232, Tampa, Florida
  - Virtus Research Consultants, LLC /ID# 217052, Wellington, Florida
  - Florida Premier Research Institute, LLC /ID# 224499, Winter Park, Florida
  - Paramount Research Solutions /ID# 218769, Alpharetta, Georgia
  - Academia of Women's Health & Endoscopic Surgery /ID# 217260, Atlanta, Georgia
  - Gyn & Fertility Specialists /ID# 223015, Atlanta, Georgia
  - Atlanta Women's Research Institute /ID# 217303, Atlanta, Georgia
  - Paramount Research Solutions - College Park /ID# 217358, College Park, Georgia
  - Duplicate_Columbus Regional Research Ins /ID# 217294, Columbus, Georgia
  - Midtown OBGYN North /ID# 222300, Columbus, Georgia
  - Innovative Women's HealthCare Solutions - Smyrna /ID# 223692, Smyrna, Georgia
  - Journey Medical Research Institute - Snellville /ID# 229774, Snellville, Georgia
  - Leavitt Womens Healthcare /ID# 217118, Idaho Falls, Idaho
  - Womens Healthcare Assoc, DBA /ID# 222153, Idaho Falls, Idaho
  - Sonora Clinical Research /ID# 222147, Meridian, Idaho
  - Asr, Llc /Id# 217094, Nampa, Idaho
  - Women's Health Care Center Of Chicago /ID# 245164, Chicago, Illinois
  - Alliance for Multispecialty Research, LLC /ID# 217226, Oak Brook, Illinois
  - The Advanced Gynecologic Surgery Institute - Park Ridge /ID# 245372, Park Ridge, Illinois
  - American Health Network of IN, LLC (Avon) /ID# 218023, Avon, Indiana
  - Investigators Research Group, LLC /ID# 222891, Brownsburg, Indiana
  - Women's Health Advantage /ID# 246580, Fort Wayne, Indiana
  - University of Iowa Hospitals and Clinics /ID# 217144, Iowa City, Iowa
  - The Iowa Clinic, PC /ID# 217351, West Des Moines, Iowa
  - GTC Research /ID# 217051, Shawnee Mission, Kansas
  - Alliance for Multispecialty Research (AMR) - Wichita West /ID# 218040, Wichita, Kansas
  - Cypress Medical Research Ctr /ID# 217093, Wichita, Kansas
  - Clinical Trials Management - Metairie /ID# 217054, Covington, Louisiana
  - Clinical Trials Management, LLC - Covington /ID# 217291, Covington, Louisiana
  - Horizon Research Group /ID# 217100, Eunice, Louisiana
  - Praetorian Pharmaceutical Research /ID# 217159, Marrero, Louisiana
  - Southern Clinical Research A /ID# 218028, Metairie, Louisiana
  - Women's Health Clinic /ID# 217205, Shreveport, Louisiana
  - SBL Special Services LLC /ID# 224899, Frederick, Maryland
  - Congressional OBGYN /ID# 245349, Rockville, Maryland
  - Continental Clinical Solutions /ID# 217053, Towson, Maryland
  - NECCR Fall River LLC /ID# 217108, Fall River, Massachusetts
  - Exordia Medical Research, Inc /ID# 217116, Fall River, Massachusetts
  - Great Lakes Research Group - Bay City /ID# 217099, Bay City, Michigan
  - Wayne State University, C.S. Mott Center /ID# 248422, Detroit, Michigan
  - Saginaw Valley Med Res Group /ID# 217296, Saginaw, Michigan
  - Center for Reproductive Medicine and Robotic Surgery /ID# 223494, St Louis, Missouri
  - Boeson Research - Great Falls /ID# 248560, Great Falls, Montana
  - Boeson Research - Missoula /ID# 248559, Missoula, Montana
  - Womens Clinic of Lincoln, P.C. /ID# 217136, Lincoln, Nebraska
  - Private practice: Dr. Rex G. Mabey JR /ID# 217134, Las Vegas, Nevada
  - Dr. Nader and Associates M.D. P.C. /ID# 223571, North Las Vegas, Nevada
  - Cooper University Hospital /ID# 227208, Camden, New Jersey
  - Jersey Shore University Medical Center /ID# 217138, Neptune City, New Jersey
  - Rutgers Robert Wood Johnson /ID# 246933, New Brunswick, New Jersey
  - Maimonides Medical Center /ID# 248493, Brooklyn, New York
  - Invision Health /ID# 218687, Buffalo, New York
  - Widewaters Gynecology /ID# 225621, East Syracuse, New York
  - Parkmed NYC /ID# 224333, New York, New York
  - Columbia Univ Medical Center /ID# 217113, New York, New York
  - New York Presbyterian Hospital Weill Cornell Medical Center /ID# 224329, New York, New York
  - Richmond OB/GYN Associates PC /ID# 224833, Staten Island, New York
  - Duplicate_PMG Research of Charlotte /ID# 217224, Charlotte, North Carolina
  - Tyron Medical Partners, PLLC /ID# 245286, Charlotte, North Carolina
  - Carolina Women's Research and Wellness Center /ID# 217133, Durham, North Carolina
  - Eastern Carolina Women's Centr /ID# 222358, New Bern, North Carolina
  - Accellacare Wilmington /ID# 217097, Wilmington, North Carolina
  - Carolina Medical Trials - Winston-Salem /ID# 223002, Winston-Salem, North Carolina
  - Unified Women's Clinical Research /ID# 217132, Winston-Salem, North Carolina
  - Unified Women's Clinical Research /ID# 218339, Winston-Salem, North Carolina
  - Clinical Inquest Center Ltd /ID# 217961, Beavercreek, Ohio
  - Neuro-Behavioral Clinical Research, Inc. /ID# 224026, Canton, Ohio
  - Seven Hills Clinical Research Group /ID# 224941, Cincinnati, Ohio
  - Duplicate_Duplicate_University Of Cincinnati Medical Center /ID# 217349, Cincinnati, Ohio
  - MetroHealth Medical Center /ID# 224392, Cleveland, Ohio
  - Central Ohio Clinical Research /ID# 217059, Columbus, Ohio
  - HWC Women's Research Center /ID# 246619, Englewood, Ohio
  - Wright State Physicians Health Center /ID# 217272, Fairborn, Ohio
  - Marion Ob/Gyn Inc. /ID# 244175, Marion, Ohio
  - Univ Hosp Landerbrook /ID# 217065, Mayfield Heights, Ohio
  - AC Clinical Research /ID# 227356, Tiffin, Ohio
  - Grube Gynecology /ID# 245132, Frackville, Pennsylvania
  - Penn State University and Milton S. Hershey Medical Center /ID# 217057, Hershey, Pennsylvania
  - University of Pennsylvania /ID# 217243, Philadelphia, Pennsylvania
  - reading Hospital /ID# 223599, Wyomissing, Pennsylvania
  - Vista Clinical Research /ID# 217151, Columbia, South Carolina
  - University Medical Group /ID# 217355, Greenville, South Carolina
  - Vitalink Research - Greenville /ID# 217075, Greenville, South Carolina
  - Duplicate_Palmetto Clinical Research /ID# 217069, Summerville, South Carolina
  - Biocentric Healthcare Research /ID# 248582, West Columbia, South Carolina
  - Chattanooga Research and Medicine /ID# 217045, Chattanooga, Tennessee
  - Research Memphis Associates, LLC /ID# 218022, Memphis, Tennessee
  - Access Clinical Trials, Inc. /ID# 217055, Nashville, Tennessee
  - DCT - HCWC, LLC dba Discovery Clinical Trials /ID# 217095, Dallas, Texas
  - Cedar Health Research /ID# 224407, Dallas, Texas
  - Duplicate_The University of Texas Southwestern Medical Center /ID# 217048, Dallas, Texas
  - Signature Gyn Services /ID# 217299, Fort Worth, Texas
  - Progressive Women's Health /ID# 248402, Friendswood, Texas
  - Willowbend Health and Wellness - Frisco /ID# 217354, Frisco, Texas
  - FMC Science, LLC - OB/GYN - Georgetown /ID# 218654, Georgetown, Texas
  - UTHealth Women's Research Program - Memorial City /ID# 217362, Houston, Texas
  - OBGYN Medical Center Associates - Medical Center Office /ID# 245346, Houston, Texas
  - Centex Studies, Inc. - Houston /ID# 217357, Houston, Texas
  - FMC Science /ID# 217047, Lampasas, Texas
  - Maximos OB/GYN /ID# 229385, League City, Texas
  - Advances in Health, Inc. /ID# 217220, Pearland, Texas
  - Clinical Trials of Texas, Inc /ID# 217039, San Antonio, Texas
  - VIP Trials /ID# 217261, San Antonio, Texas
  - Discovery Clinical Trials-San Antonio /ID# 218547, San Antonio, Texas
  - Center of Reproductive Medicine /ID# 217241, Webster, Texas
  - Corner Canyon Obstetrics and G /ID# 217289, Draper, Utah
  - Duplicate_Physicians Research Options /ID# 217302, Pleasant Grove, Utah
  - Highland Clinical Research /ID# 224052, Salt Lake City, Utah
  - Health Research of Hampton Roads, Inc. (HRHR) /ID# 217063, Newport News, Virginia
  - Clinical Research Partners /ID# 217359, North Chesterfield, Virginia
  - Virginia Women's Health Associates /ID# 227677, Reston, Virginia
  - Clinical Trials Virginia, Inc. /ID# 217222, Richmond, Virginia
  - Clinical Research Partners LLC - Richmond Forest Ave /ID# 217149, Richmond, Virginia
  - Tidewater Clinical Research /ID# 217152, Virginia Beach, Virginia
  - Seattle Clinical Research Center /ID# 217117, Seattle, Washington
  - North Spokane Women's Health /ID# 217356, Spokane, Washington
- Puerto Rico (3):
  - Advanced Medical Concepts. PSC /ID# 221337, Cidra
  - Henry A. Rodriguez Ginorio, MD /ID# 217233, San Juan
  - School of Medicine University of Puerto Rico-Medical Science Campus /ID# 217235, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M18-969